CLINICAL TRIAL: NCT03093142
Title: The Treatment Effectiveness of Combined tDCs and Neurofeedback (NF) for Patients With Cognitive Deficits After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kowloon Hospital, Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Marko Chan, Principal Investigator, Kowloon Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KowloonH
Record Dates: First submitted 2017-03-01; First posted 2017-03-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Cognitive Impairment
Keywords: transcranial direct current stimulation (tDCs); neurofeedback
MeSH Terms: conditions — Stroke; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation; Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS & neurofeedback (Experimental): 30 minutes tDCS & 30 minutes neurofeedback
  Interventions: Device: tDCS & neurofeedback
- real neurofeedback (Active Comparator): 30 minutes real neurofeedback.
  Interventions: Device: neurofeedback
- sham neurofeedback (Sham Comparator): 30 minutes sham neurofeedback.
  Interventions: Device: sham neurofeedback

INTERVENTIONS:
Device: tDCS & neurofeedback — tDCs and neurofeedback
  Arms: tDCS & neurofeedback
Device: neurofeedback — Neurofeedback
  Arms: real neurofeedback
Device: sham neurofeedback — sham neurofeedback
  Arms: sham neurofeedback

SUMMARY:
This is a double blinded, randomized control trial with a pretest-posttest control and interventional groups design. Both the assessor and participants are blinded to all assessments and evaluations. All patients with subacute stroke undergo in-patient or out-patient rehabilitation are screened initially by a series of screening test. Suitable patients are assigned randomly to 3 groups respectively. Group 1 is the combined transcranial direct current stimulation (tDCS) and neurofeedback group. Group 2 is the neurofeedback group. Group 3 is the control group with sham neurofeedback training.

DETAILED DESCRIPTION:
Treatment sessions for all three groups are conducted by the investigators who has training in neurofeedback and transcranial direct current stimulation (tDCs). Each participant performed 10 training sessions on different days. Sessions were conducted 3-5 times a week The tDCS + neurofeedback group will carry out 30 minutes tDCS and 30 minutes neurofeedback training.

The real neurofeedback group will carry out 30 minutes neurofeedback training. The sham neurofeedback group will conduct the 30 minutes sham neurofeedback training.

ELIGIBILITY:
Inclusion Criteria:

1. First or second stroke (haemorrhagic or ischaemic) confirmed by computer axial tomography scan or magnetic resonance imaging
2. Below 16 th percentile cut off in Hong Kong Montreal - Cognitive Assessment (HK - MoCA) (range from 17-25/30).
3. Less than twelve months since onset of stroke at study entry
4. Able to follow simple command

Exclusion Criteria:

1. Patients with severe dysphasia (either expressive or comprehensive) which restricts communication;
2. History of other neurological disease, psychiatric disorder, or alcoholism;
3. Significant impairment in visual or auditory function
4. Any additional medical or psychological condition that would affect their ability to comply with the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change score in Trail Making Test A & B from baseline | One day before the treatment , up to 4 weeks, up to 16 weeks
  Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.

SECONDARY OUTCOMES:
Change score in Functional Independence Measure (FIM) from baseline | One day before the treatment , up to 4 weeks, up to 16 weeks
  The Functional Independence Measure instrument is a basic indicator of patient disability. FIM is used to track the changes in the functional ability of a patient during an episode of hospital rehabilitation care.
Change score in Stroke Adapted 30 item version of the Sickness Impact Profile (SA - SIP 30) | One day before the treatment , up to 4 weeks, up to 16 weeks
  SA-SIP 30 assesses quality of life in patients who have sustained a stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Marko Chan, PhDCandidate, Principal Investigator — Community Rehabilitation Service Supoort Centre
Locations (1):
- Community Rehabilitation Service Support Centre, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No